CLINICAL TRIAL: NCT02336230
Title: A Single-arm, Prospective Study of Remestemcel-L, Ex-vivo Culture-Expanded Adult Human Mesenchymal Stromal Cells, for the Treatment of Pediatric Patients Who Have Failed to Respond to Steroid Treatment for Acute GVHD
Brief Title: A Prospective Study of Remestemcel-L, Ex-vivo Cultured Adult Human Mesenchymal Stromal Cells, for the Treatment of Pediatric Participants Who Have Failed to Respond to Steroid Treatment for Acute Graft-Versus-Host Disease (aGVHD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mesoblast, Inc. (Industry)
Collaborators: Quintiles, Inc. (Industry)
Responsible Party: Sponsor
Organization: Mesoblast, Ltd. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MSB-GVHD001
Record Dates: First submitted 2014-12-30; First posted 2015-01-12 (Estimated); Results first posted 2022-03-17 (Actual); Last update posted 2022-03-17 (Actual); Status verified 2022-02

CONDITIONS: Grade B aGVHD; Grade C aGVHD; Grade D aGVHD
Keywords: GVHD
MeSH Terms: interventions — remestemcel-l

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Remestemcel-L 2×10^6 MSCs/kg (Experimental): Participants were treated with intravenous (IV) remestemcel-L at a dose of 2×10^6 mesenchymal stromal cells (MSCs)/kilogram (kg) actual body weight at Screening, twice per week, for each of 4 consecutive weeks (initial therapy) given at least 3 days apart and no more than 5 days apart for any infusion. Eligible participants received an additional once per week infusion, for each of 4 consecutive weeks (continued therapy) of remestemcel-L and twice per week infusions, for each of 4 consecutive weeks (aGVHD flare therapy) of remestemcel-L at the same initial therapy dose of 2×10^6 MSCs/kg actual body weight at Screening.
  Interventions: Drug: remestemcel-L

INTERVENTIONS:
Drug: remestemcel-L — Participants were treated with IV remestemcel-L at a dose of 2 x 10^6 MSC/kg (actual body weight at screening) twice per week for each of 4 consecutive weeks. Infusions were administered at least 3 days apart and no more than 5 days apart for any infusion.

SUMMARY:
The study plans to treat at least 60 pediatric participants, male and female, between the ages of 2 months and 17 years inclusive with aGVHD following allogeneic hematopoietic stem cell transplant (HSCT) that has failed to respond to treatment with systemic corticosteroid therapy. Participants may have Grades C and D aGVHD involving the skin, liver and/or gastrointestinal (GI) tract or Grade B aGVHD involving the liver and/or GI tract, with or without concomitant skin disease.

DETAILED DESCRIPTION:
Remestemcel-L will be evaluated in pediatric participants with aGVHD following allogeneic HSCT that has failed to respond to treatment with systemic corticosteroid therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Participant is diagnosed with Grade B-D acute GVHD requiring corticosteroid systemic therapy. The participant may have Grade C or D aGVHD involving the skin, liver, and/or GI tract or may have Grade B aGVHD involving the liver and/or GI tract, with or without concomitant skin disease. Acute GVHD is defined as the presence of skin rash and/or persistent nausea, vomiting, and/or diarrhea and/or cholestasis presenting in a context in which aGVHD is likely to occur and where other etiologies such as drug rash, enteric infection, or hepatotoxic syndromes are unlikely or have been ruled out.
2. Participant has failed to respond to steroid treatment, with failure to respond defined as any Grade B-D [International Bone Marrow Transplant Registry (IBMTR) grading] aGVHD that shows progression within 3 days, or no improvement within 7 days of consecutive treatment with 2 mg/kg/day methylprednisolone or equivalent.
3. Participant must be able to be treated with remestemcel-L within 4 days of signing of informed consent.
4. Participants who have had persistent GI GVHD manifested by diarrhea with stool volume < 500 mL/kg/day (for participants >50 kg) or <30 mL/kg/day (for participants ≤50 kg). See GVHD Organ Severity Criteria (Table 2) for values in mL/m^2. In the absence of nausea or vomiting, participants could have been considered to have Grade B GVHD if:

   1. other causes of diarrhea had been ruled out (eg, Clostridium difficile, adenovirus or cytomegalovirus [CMV] infection, or oral magnesium administration), and if
   2. the low stool volume reflected the effects of fasting, narcotics, or antidiarrheal medications.
5. Participant must have adequate renal function as defined by a calculated creatinine clearance of >30 mL/min per 1.73 m^2. For participants 1 to 18 years of age, creatinine clearance is calculated using the Bedside Schwartz equation:

   Glomerular filtration rate (GFR, in mL/min per 1.73 m^2) = (0.413 * height [cm])/serum creatinine (mg/dL)

   For participants younger than 1 year of age, renal function is determined using the Schwartz equation adjusted for this age group:

   Creatinine clearance (mL/min per 1.73 m^2= (height [cm] x 0.45)/ (serum creatinine [mg/dL]).
6. Participant has a minimum Karnofsky/Lansky Performance Level of at least 30 at the time of study entry.
7. Participant (or legal representative where appropriate) must be capable of providing written informed consent.
8. Female participants of childbearing potential (≥10 years of age) are required to use a medically accepted method of contraception and to agree to continue use of this method for the duration of the study and for the follow-up time period. Acceptable methods of contraception include abstinence, barrier method with spermicide, intrauterine device (IUD), or steroidal contraceptive (oral, transdermal, implanted, and injected) in conjunction with a barrier method.
9. Male participants with partners of childbearing potential must agree to use adequate contraception (barrier method or abstinence) during the study, including the follow-up time period.
10. The participant must be willing and able to comply with study requirements, remain at the clinic, and return to the clinic for the follow-up evaluation during the study period, as specified in this protocol.

Exclusion Criteria:

1. Participant has Grade B aGvHD with skin-only involvement.
2. Participant has received any second line therapy to treat aGVHD prior to screening.
3. Participant has received systemic agents other than steroids and prophylactic agents for primary treatment of aGVHD.
4. Participant shows evidence of diffuse alveolar hemorrhage or other active pulmonary disease, which is likely to require more than 2L of oxygen via face mask, or an estimated fractional inspired oxygen concentration (FiO2) of 28% via other delivery methods in order to sustain an O2 saturation of 92%.
5. Participant has any underlying or current medical or psychiatric condition that, in the opinion of the Investigator, would interfere with the evaluation of the participant including but not limited to uncontrolled infection, heart failure, or pulmonary hypertension.
6. Participant has received any stem cell agents (other than hematopoietic graft) during study participation or within 30 days prior to study entry. Previous use of irradiated granulocytes within 30 days is permitted.
7. Participant has received an HSCT transplant for a solid tumor disease.
8. Participant has had prior treatment with mesenchymal stem cells (MSCs), including remestemcel-L.
9. Participant shows evidence of severe (required treatment) hepatic veno-occlusive disease (VOD) or sinusoidal obstruction at screening.
10. Participant had positive laboratory test results indicating infection with the human immunodeficiency virus (HIV) at any time and/or active hepatitis B or C virus infection within 3 months prior to screening.
11. Participant shows evidence of encephalopathy, as defined by a change in mental status since the onset of aGVHD.
12. Participant is a female who is pregnant, lactating, or is planning a pregnancy during study participation, or in the follow-up period.
13. Participant currently being treated for a solid tumor malignancy.
14. Participant has participated in any interventional clinical trial for an aGVHD therapeutic agent. However, in exceptional cases, experimental agents may have been administered to enrolled participants at the Investigator's discretion.
15. Participant has participated or is currently participating in any autologous and allogeneic stem cell or gene therapy study for the treatment of aGVHD. Participants participating in investigative protocols aimed at modification of the transplant graft (such as T-cell depletion) or aimed at modification of the conditioning regimen are allowed in the study.
16. Participant has a known hypersensitivity to dimethyl sulfoxide (DMSO) or to murine, porcine, or bovine proteins.

Ages: 2 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 55 (Actual)
Dates: Start 2015-06-04 (Actual); Primary Completion 2018-04-09 (Actual); Study Completion 2018-04-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher James, Study Director — Mesoblast, Inc.
Locations (20):
- United States (20):
  - Children's Hospital Los Angeles, Los Angeles, California
  - Children's Hospital of Orange County, Orange, California
  - University of California at San Francisco, San Francisco, California
  - Children's Hospital Colorado Center for Cancer/Blood Disorders, Aurora, Colorado
  - Alfred I. DuPont Hospital for Children of the Nemours Foundation, Wilmington, Delaware
  - Miami Children's Research Institute, Miami, Florida
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Children's Hospital of Michigan, Detroit, Michigan
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Washington University, St Louis, Missouri
  - Columbia University Medical Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Albert Einstein College of Medicine, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Oregon University, Portland, Oregon
  - Medical University of South Carolina, Charleston, South Carolina
  - Texas Transplant Institute, San Antonio, Texas
  - Virginia Commonwealth University, Richmond, Virginia
  - Fred Hutchinson Cancer Research, Seattle, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kurtzberg J, Abdel-Azim H, Carpenter P, Chaudhury S, Horn B, Mahadeo K, Nemecek E, Neudorf S, Prasad V, Prockop S, Quigg T, Satwani P, Cheng A, Burke E, Hayes J, Skerrett D; MSB-GVHD001/002 Study Group. A Phase 3, Single-Arm, Prospective Study of Remestemcel-L, Ex Vivo Culture-Expanded Adult Human Mesenchymal Stromal Cells for the Treatment of Pediatric Patients Who Failed to Respond to Steroid Treatment for Acute Graft-versus-Host Disease. Biol Blood Marrow Transplant. 2020 May;26(5):845-854. doi: 10.1016/j.bbmt.2020.01.018. Epub 2020 Feb 1. PMID 32018062

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Remestemcel-L 2×10^6 MSCs/kg
Started | 55
Full Analysis Set (FAS) (The FAS included all participants who provided informed consent, were screened, and were found eligible to enter the study.) | 55
Safety Analysis Population (The Safety Analysis Population included all participants who signed the informed consent form and received at least 1 dose of remestemcel-L.) | 54
Completed | 42
Not Completed | 13
Not completed — Adverse Event | 1
Not completed — Withdrawal of consent | 1
Not completed — Death | 9
Not completed — Dose not received due to shipping delay | 1
Not completed — Discontinuation of MSC infusion | 1

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) included all participants who provided informed consent, were screened, and were found eligible to enter the study.
Groups:
- Remestemcel-L 2×10^6 MSCs/kg: Participants were treated with IV remestemcel-L at a dose of 2×10^6 MSCs/kg actual body weight at Screening, twice per week, for each of 4 consecutive weeks (initial therapy) given at least 3 days apart and no more than 5 days apart for any infusion. Eligible participants received an additional once per week infusion, for each of 4 consecutive weeks (continued therapy) of remestemcel-L and twice per week infusions, for each of 4 consecutive weeks (aGVHD flare therapy) of remestemcel-L at the same initial therapy dose of 2×10^6 MSCs/kg actual body weight at Screening.
Arm/Group | Remestemcel-L 2×10^6 MSCs/kg
Number analyzed (Participants) | 55
Age, Continuous [Mean (Standard Deviation); unit: years] | 7.3 (5.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 35
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 18
  Not Hispanic or Latino | 36
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 8
  White | 31
  More than one race | 10
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR) at Day 28 Post Initiation of Therapy
Description: ORR was defined as the percentage of participants who had achieved overall response. Overall response was defined as complete response (CR) plus partial response (PR) as per aGVHD response criteria. CR was defined as resolution of aGVHD in all involved organs. PR was defined as organ improvement of at least 1 stage without worsening of any other organ.
Time Frame: Day 28
Population: FAS included all participants who provided informed consent, were screened, and were found eligible to enter the study.
Measure: Number; unit: percentage of participants
Arm/Group | Remestemcel-L 2×10^6 MSCs/kg
Number analyzed (Participants) | 55
percentage of participants | 69.1
Statistical Analysis 1: Comparison: Remestemcel-L 2×10^6 MSCs/kg; Test type: Other; p = 0.0003, Binomial Distribution — P-value was calculated from the binomial distribution under the assumption of a 0.45 success rate for the null hypothesis

2. Secondary Outcome: Overall Survival (OS) Rate at Day 100 Post Initiation of Therapy
Description: Overall survival rate was defined as percentage of participants who survived. OS was defined as the time to death from the start of drug therapy.
Time Frame: Day 100
Population: FAS included all participants who provided informed consent, were screened, and were found eligible to enter the study.
Measure: Number; unit: percentage of participants
Arm/Group | Remestemcel-L 2×10^6 MSCs/kg
Number analyzed (Participants) | 55
percentage of participants | 74.5

3. Secondary Outcome: OS Rate at Day 100 Post Initiation of Therapy, Stratified by Responder Status at Day 28
Description: as for outcome 2
Time Frame: Day 100
Population: FAS included all participants who provided informed consent, were screened, and were found eligible to enter the study. Number analyzed is the number of participants with data available for given category.
Measure: Number; unit: percentage of participants
Arm/Group | Remestemcel-L 2×10^6 MSCs/kg
Number analyzed (Participants) | 55
percentage of participants
  Responders: number analyzed (Participants) | 38
  Responders | 86.8
  Non- Responders: number analyzed (Participants) | 17
  Non- Responders | 47.1
Statistical Analysis 1: Comparison: Remestemcel-L 2×10^6 MSCs/kg; Test type: Other; p = 0.0032, CHM test — P-value was from a Cochran-Mantel-Haenszel (CMH) test stratified by baseline aGVHD grade

4. Secondary Outcome: OS Rate at Day 100 Post Initiation of Therapy, Stratified by Baseline aGVHD Grade
Description: OS rate was defined as percentage of participants who survived. OS was defined as the time to death from the start of drug therapy. Maximum severity of acute GVHD was assessed by using International Bone Marrow Transplant Registry (IBMTR) index. The severity index was defined as: Grade A (skin Stage 1: extent of rash <25%); Grade B (skin Stage 2: extent of rash 25 to 50% or liver Stage 1 to 2: total bilirubin 34 to 102 micromoles per liter [mcmol/L] or intestinal tract Stage 1 to 2: volume of diarrhea 550 to 1500 milliliters per day [mL/day]); Grade C (skin Stage 3: extent of rash > 50% or liver Stage 3: total bilirubin 103 to 255 mcmol/L or intestinal tract Stage 3: volume of diarrhea >1500 mL/day); Grade D (skin Stage 4: extent of rash bullae or liver Stage 4: total bilirubin >255 or intestinal tract Stage 4: volume of diarrhea severe pain and ileus).
Time Frame: Day 100
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Remestemcel-L 2×10^6 MSCs/kg
Number analyzed (Participants) | 55
percentage of participants
  Grade A: number analyzed (Participants) | 0
  Grade B: number analyzed (Participants) | 6
  Grade B | 50.0 [11.81 to 88.19]
  Grade C: number analyzed (Participants) | 23
  Grade C | 82.6 [61.22 to 95.05]
  Grade D: number analyzed (Participants) | 26
  Grade D | 73.1 [52.21 to 88.43]

5. Secondary Outcome: OS Rate at Day 100 Post Initiation of Therapy, Stratified by Organ Involvement
Description: OS rate was defined as percentage of participants who survived. OS was defined as the time to death from the start of drug therapy. The data was summarized for organ involvement: skin only, lower GI only, and multi-organ.
Time Frame: Day 100
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Remestemcel-L 2×10^6 MSCs/kg
Number analyzed (Participants) | 55
percentage of participants
  Skin Only: number analyzed (Participants) | 14
  Skin Only | 78.6
  Lower GI Only: number analyzed (Participants) | 21
  Lower GI Only | 76.2
  Multi-organ (Any Combination): number analyzed (Participants) | 20
  Multi-organ (Any Combination) | 70.0

6. Secondary Outcome: OR Rate at Day 56 and 100 Post Initiation of Therapy
Description: OR rate was defined as the percentage of participants who had achieved overall response. Overall response was defined as CR plus PR as per aGVHD response criteria. CR was defined as resolution of aGVHD in all involved organs. PR was defined as organ improvement of at least 1 stage without worsening of any other organ.
Time Frame: Day 56 and Day 100
Population: FAS included all participants who provided informed consent, were screened, and were found eligible to enter the study.
Measure: Number; unit: percentage of participants
Arm/Group | Remestemcel-L 2×10^6 MSCs/kg
Number analyzed (Participants) | 55
percentage of participants
  Day 56 | 58.2
  Day 100 | 69.1

ADVERSE EVENTS:
Time Frame: From Baseline through 100 days of follow up
Description: All-cause Mortality: FAS included all participants who provided informed consent, were screened, and were found eligible to enter the study. Serious and Other (Non-serious) AEs: Safety Analysis Population included all participants who signed the informed consent form and received at least 1 dose of remestemcel-L.
Arm/Group | Remestemcel-L 2×10^6 MSCs/kg
All-Cause Mortality (participants affected / at risk) | 13/55
Serious Adverse Events (participants affected / at risk) | 35/54
Other Adverse Events (participants affected / at risk) | 52/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Remestemcel-L 2×10^6 MSCs/kg (N=54)
Haemolytic uraemic syndrome (Blood and lymphatic system disorders) | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Haemolysis (Blood and lymphatic system disorders) | 1
Pancytopenia (Blood and lymphatic system disorders) | 1
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 1
Cardiac arrest (Cardiac disorders) | 1
Cardiac failure (Cardiac disorders) | 1
Pericardial effusion (Cardiac disorders) | 1
Pneumatosis intestinalis (Gastrointestinal disorders) | 4
Abdominal pain (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Jejunal perforation (Gastrointestinal disorders) | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Pyrexia (General disorders) | 5
Multiple organ dysfunction syndrome (General disorders) | 5
Asthenia (General disorders) | 1
Acute graft versus host disease (Immune system disorders) | 3
Graft versus host disease in skin (Immune system disorders) | 2
Graft versus host disease (Immune system disorders) | 1
Staphylococcal infection (Infections and infestations) | 3
BK virus infection (Infections and infestations) | 2
Escherichia urinary tract infection (Infections and infestations) | 2
Human herpesvirus 6 infection (Infections and infestations) | 2
Pneumonia (Infections and infestations) | 2
Sepsis (Infections and infestations) | 2
Staphylococcal bacteraemia (Infections and infestations) | 2
Adenovirus infection (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Clostridium difficile infection (Infections and infestations) | 1
Enterococcal infection (Infections and infestations) | 1
Epstein-Barr viraemia (Infections and infestations) | 1
Fungaemia (Infections and infestations) | 1
Fungal infection (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Lactobacillus infection (Infections and infestations) | 1
Rotavirus infection (Infections and infestations) | 1
Staphylococcal sepsis (Infections and infestations) | 1
Platelet count decreased (Investigations) | 1
White blood cell count decreased (Investigations) | 1
Dehydration (Metabolism and nutrition disorders) | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 1
Hypermetabolism (Metabolism and nutrition disorders) | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 1
Acute myeloid leukaemia recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Acute megakaryocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 2
Somnolence (Nervous system disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 1
Cystitis haemorrhagic (Renal and urinary disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 5
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 2
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1
Capillary leak syndrome (Vascular disorders) | 1
Hypertensive crisis (Vascular disorders) | 1
Hypovolaemic shock (Vascular disorders) | 1
Peripheral ischaemia (Vascular disorders) | 1
Shock haemorrhagic (Vascular disorders) | 1
Venoocclusive disease (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Remestemcel-L 2×10^6 MSCs/kg (N=54)
Anaemia (Blood and lymphatic system disorders) | 4
Neutropenia (Blood and lymphatic system disorders) | 3
Sinus tachycardia (Cardiac disorders) | 5
Pericardial effusion (Cardiac disorders) | 3
Tachycardia (Cardiac disorders) | 3
Adrenal insufficiency (Endocrine disorders) | 5
Cushingoid (Endocrine disorders) | 5
Abdominal pain (Gastrointestinal disorders) | 10
Vomiting (Gastrointestinal disorders) | 9
Diarrhoea (Gastrointestinal disorders) | 6
Abdominal distension (Gastrointestinal disorders) | 4
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 4
Haematochezia (Gastrointestinal disorders) | 4
Constipation (Gastrointestinal disorders) | 3
Flatulence (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 3
Pyrexia (General disorders) | 13
Oedema peripheral (General disorders) | 7
Generalised oedema (General disorders) | 3
Hyperbilirubinaemia (Hepatobiliary disorders) | 3
Chronic graft versus host disease (Immune system disorders) | 6
Hypogammaglobulinaemia (Immune system disorders) | 6
Graft versus host disease in skin (Immune system disorders) | 3
Adenovirus infection (Infections and infestations) | 10
Epstein-Barr viraemia (Infections and infestations) | 7
BK virus infection (Infections and infestations) | 5
Epstein-Barr virus infection (Infections and infestations) | 4
Urinary tract infection (Infections and infestations) | 4
Cytomegalovirus infection (Infections and infestations) | 3
Oral candidiasis (Infections and infestations) | 3
Pneumonia fungal (Infections and infestations) | 3
Allergic transfusion reaction (Injury, poisoning and procedural complications) | 3
Transaminases increased (Investigations) | 5
Alanine aminotransferase increased (Investigations) | 4
Blood creatinine increased (Investigations) | 3
Electrocardiogram QT prolonged (Investigations) | 3
Hyperglycaemia (Metabolism and nutrition disorders) | 7
Hypokalaemia (Metabolism and nutrition disorders) | 7
Hypomagnesaemia (Metabolism and nutrition disorders) | 6
Hyponatraemia (Metabolism and nutrition disorders) | 5
Hypophosphataemia (Metabolism and nutrition disorders) | 4
Hyperkalaemia (Metabolism and nutrition disorders) | 3
Hypernatraemia (Metabolism and nutrition disorders) | 3
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 3
Hypoalbuminaemia (Metabolism and nutrition disorders) | 3
Malnutrition (Metabolism and nutrition disorders) | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 8
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4
Joint swelling (Musculoskeletal and connective tissue disorders) | 3
Headache (Nervous system disorders) | 4
Tremor (Nervous system disorders) | 3
Agitation (Psychiatric disorders) | 4
Anxiety (Psychiatric disorders) | 3
Insomnia (Psychiatric disorders) | 3
Cystitis haemorrhagic (Renal and urinary disorders) | 5
Acute kidney injury (Renal and urinary disorders) | 4
Dysuria (Renal and urinary disorders) | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 7
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3
Dry skin (Skin and subcutaneous tissue disorders) | 3
Rash papular (Skin and subcutaneous tissue disorders) | 3
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 3
Skin ulcer (Skin and subcutaneous tissue disorders) | 3
Hypertension (Vascular disorders) | 10
Hypotension (Vascular disorders) | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publications (abstracts, posters or presentations) must be presented to the Publication Steering Committee for review prior to submission or public display and are not allowed prior to the publication of the primary manuscript, or eighteen (18) months from the conclusion of the Study. PI shall provide Sponsor a copy of any proposed public disclosure at least 30 days prior to submission. Sponsor may ask PI to delay the disclosure for a maximum of 60 days to file proprietary protection.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-08): https://cdn.clinicaltrials.gov/large-docs/30/NCT02336230/Prot_SAP_000.pdf